CLINICAL TRIAL: NCT02396498
Title: S-1 With Cisplatin Intravenous Chemotherapy Versus S-1 Plus Cisplatin Hyperthermic Intraperitoneal Chemotherapy in Stage Ⅲ Patients After D2 Gastrectomy：a Randomized Controlled Study
Brief Title: SP Intravenous Chemotherapy Versus SP by HIPEC in Stage Ⅲ Patients After D2 Gastrectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TDCCC005
Record Dates: First submitted 2014-11-11; First posted 2015-03-24 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Stage Ⅲ Gastric Cancer
MeSH Terms: interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D2 radical gastrectomy+Systemic chemotherapy (Placebo Comparator): 8 cycles of systemic chemotherapy were performed for stage Ⅲ patients after D2 gastrectomy .Systemic chemotherapy(SP): Cisplatin: 60mg/m^2, d1 , Intravenous infusion, every 3 weeks. S-1: 40-60mg/m^2 bid, days 1-14, every 3 weeks .Subjects should be given maximum 8 cycles, or progression/intolerance.
- D2 radical gastrectomy+HIPEC (Experimental): 8 cycles of hyperthermic intraperitoneal chemotherapy (cisplatin) and S-1(oral) were performed after D2 radical gastrectomy. HIPEC was conducted in d1 and d3: Normal saline 2000ml-5000ml, Cisplatin 60mg/m^2, 43°C, 60min. every 3 weeks. S-1: 40-60mg/m^2 bid, days 1-14, every 3 weeks.Subjects should be given maximum 8 cycles, or progression/intolerance.
  Interventions: Drug: HIPEC

INTERVENTIONS:
Drug: HIPEC — Using cisplatin in HIPEC plus oral S-1
  Other Names: hyperthermic intraperitoneal chemoperfusion
  Arms: D2 radical gastrectomy+HIPEC

SUMMARY:
The study is designed to assess the safety and efficacy of S-1 plus cisplatin hyperthermic intraperitoneal chemotherapy in stage Ⅲ patients after D2 gastrectomy

DETAILED DESCRIPTION:
The study is a randomized clinical trial，and subjects wuill be assigned two arms: SP Intravenous Chemotherapy or SP by HIPEC .After 8 cycles treatment,we assess the safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* 18 ≤ age ≤ 70 years old
* Histologically diagnosed as stageⅢ gastric adenocarcinoma，and perform D2 radical gastrectomy，as well as have not received any Anti-tumor therapy：chemotherapy,biological treatment or molecular targeted therapy , etc.
* The Eastern Cooperative Oncology Group (ECOG) status ≤ 2
* Having given written informed consent prior to any procedure related to the study
* Expected survival time ≥3 months

Exclusion Criteria:

* History of severe hypersensitivity reactions to the ingredients of S-1 or Cisplatin
* Hemoglobin<90g/L
* Inadequate hematopoietic function which is defined as below:

  * white blood cell (WBC) less than 3,500/mm^3
  * absolute neutrophil count (ANC) less than 1,500/mm^3
  * platelets less than 80,000/mm^3
* Inadequate hepatic or renal function which is defined as below:

  * serum bilirubin greater than 2 times the upper limit of normal range
  * alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 2.5 times the ULN if no demonstrable liver metastases or greater than 5 times the ULN in the presence of liver metastases
  * blood creatinine level greater than 1.5 times ULN,Creatinine clearance<60ml/min
* Receiving a concomitant treatment with other fluoropyrimidine drug or flucytosine drug
* Women who is pregnant or lactating or fertile women of child-bearing potential unless using a reliable and appropriate contraceptive method throughout the treatment period (Including male)
* Psychiatric disorder or symptom that makes participation of the patient difficult
* Myocardial infarction, existing serious or unstable angina, and patients with cardiac insufficiency in 6 months
* Severe complication(s), e.g., paresis of intestines, ileus, radiographically confirmed interstitial pneumonitis or pulmonary fibrosis, glomerulonephritis ,renal failure, poorly-controlled diabetes
* Known DPD deficiency
* Participate in other clinical trial before the start of this trial
* Patient compliance is bad or researchers believe that patients are not suitable for this treatment
* Known to have active hepatitis patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
DFS: Disease-Free Survival | 2 years
  from the date of random to the date of recurrence or death for disease progression.

SECONDARY OUTCOMES:
OS: Overall Survival | 5 years
  From the date of random to the date of death or to the end of follow-up
The quality of life | 6 months
  The subjects should finish the quality of life scale by themselves before treament in every cycle.
Safety as measured by Adverse Events and Serious Adverse events In the process of the total treatment according CTCAE4.0 | 6 months
  record and collect subjects' AE and SAE In the process of the total treatment according CTCAE4.0

CONTACTS AND LOCATIONS:
Overall Officials: Helong Zhang, Professor, Principal Investigator — Tang-Du Hospital
Locations (1):
- IEC of Insititution for National Drug Clinical Trials,Tangdu Hospital,Fourth Military Medical University, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Liu L, Sun L, Zhang N, Liao CG, Su H, Min J, Song Y, Yang X, Huang X, Chen D, Chen Y, Zhang HW, Zhang H. A novel method of bedside hyperthermic intraperitoneal chemotherapy as adjuvant therapy for stage-III gastric cancer. Int J Hyperthermia. 2022;39(1):239-245. doi: 10.1080/02656736.2022.2028018. PMID 35100917